CLINICAL TRIAL: NCT01220557
Title: Prospective Randomized Trial for the Evaluation of a Treatment and Education Programme for Type 1 Diabetic Patients (PRIMAS)
Brief Title: Evaluation of a Treatment and Education Programme for Type 1 Diabetic Patients (PRIMAS)
Acronym: PRIMAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Forschungsinstitut der Diabetes Akademie Mergentheim (Other)
Responsible Party: Principal Investigator, Norbert Hermanns, PhD, Forschungsinstitut der Diabetes Akademie Mergentheim
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NH062010
Record Dates: First submitted 2010-10-12; First posted 2010-10-14 (Estimated); Results first posted 2014-08-26 (Estimated); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Type 1 Diabetes
Keywords: Diabetes mellitus, education, self management
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — thymidine 5'-triphosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PRIMAS group (Experimental): PRIMAS is a newly developed treatment and education programme for type 1 diabetic patients. It consists of 12 lessons (duration 90 minutes each), slides for diabetes educators and patient material
  Interventions: Behavioral: PRIMAS
- Control group (Active Comparator): The German DTTP (Diabetes Teaching and Treatment Programme) - The German ZI Program - is an established treatment and education programme for intensified insulin treatment consisting of 12 lessons (90 minutes duration each). Flipchart for diabetes educators and patient material.
  Interventions: Behavioral: DTTP

INTERVENTIONS:
Behavioral: PRIMAS — PRIMAS is a newly developed treatment and education programme for type 1 diabetic patients. It consists of 12 lessons (duration 90 minutes each), slides for diabetes educators and patient material
  Arms: PRIMAS group
Behavioral: DTTP — The German DTTP (Diabetes Teaching and Treatment Programme) - The German ZI Program - is an established treatment and education programme for intensified insulin treatment consisting of 12 lessons (90 minutes duration each). Flipchart for diabetes educators and patient material.
  Other Names: The German Diabetes Teaching and Treatment Programme; ZI Treatment and Education Program for intensified insulin theapy
  Arms: Control group

SUMMARY:
This study is a randomized prospective trial with 6-month follow up. A non-inferiority hypothesis is tested. A new developed treatment and education programme for type 1 diabetic patients (PRIMAS) will be tested compared to an established treatment and education programme (German DTTP). Primary outcome variable is glycemic control at 6-month follow up. Secondary outcome variables are: diabetes knowledge, diabetes related distress, depressive symptoms, diabetes self-efficacy, self-care behavior, attitudes towards diabetes and insulin treatment, hypoglycemia awareness.

DETAILED DESCRIPTION:
Both programmes consists of 12 lessons with a length of 90 minutes. Eligible type 1 diabetic patients in a diabetologist practice are pooled and randomised either to the new developed PRIMAS programme or to an established education programme for type 1 diabetic patients (DTTP - Treatment and education programme for intensified insulin treatment) as an active comparator.

ELIGIBILITY:
Inclusion criteria:

type 1 diabetes, diabetes duration > 4 weeks, age 18 - 75 years, BMI 20 - 40 kg/m², A1c 7 - 13 %, ability to understand, speak and write German language, written informed consent.

Exclusion criteria:

current treatment of psychological or psychiatric disorder, dementia or severe cognitive impairment, severe organic disease (e.g. terminal renal disease, cancer with poor prognosis), preventing a regular participation in the training course, pregnancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2010-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Hermanns, PhD, Principal Investigator — Forschungsinstitut der Diabetes Akademie Mergentheim (FIDAM GmbH)

REFERENCES:
- [Result] Hermanns N, Kulzer B, Ehrmann D, Bergis-Jurgan N, Haak T. The effect of a diabetes education programme (PRIMAS) for people with type 1 diabetes: results of a randomized trial. Diabetes Res Clin Pract. 2013 Dec;102(3):149-57. doi: 10.1016/j.diabres.2013.10.009. Epub 2013 Oct 9. PMID 24210673

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participants were recruited in 23 outpatient study centres, which were located all over Germany. A study centre was defined as a medical practice run by a diabetologist and a diabetes educator or diabetes nurse.
Period: Overall Study
Arm/Group | PRIMAS Group | Control Group
Started | 81 | 79
Completed | 75 (per protocol analysis including patients which participated in at least 6 out of 12 lessons.) | 74 (per protocol analysis including patients which participated in at least 6 out of 12 lessons.)
Not Completed | 6 | 5
Not completed — Lost to Follow-up | 5 | 3
Not completed — attended less than 6 lessons | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PRIMAS Group | Control Group | Total
Number analyzed (Participants) | 81 | 79 | 160
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 74 | 77 | 151
  >=65 years | 7 | 2 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (13.8) | 45.1 (13.4) | 45.5 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 39 | 70
  Male | 50 | 40 | 90
Region of Enrollment [Number; unit: participants]
  Germany | 81 | 79 | 160

OUTCOME MEASURES:

1. Primary Outcome: Changes in Glycemic Control Measured by A1c
Description: Difference between baseline A1c and A1c at 6 month follow up. Equivalent effect on glycemic control measured by A1c (non-inferiority). In case of-non-inferiority test of superiority.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: Changes in A1c in percentage points
Arm/Group | PRIMAS Group | Control Group
Number analyzed (Participants) | 75 | 74
Changes in A1c in percentage points | -0.4 (1.0) | 0.0 (0.6)

2. Secondary Outcome: Diabetes Knowledge
Description: To assess knowledge among insulin-treated diabetes patients, participants completed a new developed 11-item diabetes knowledge score. Each item had to be answered by selecting the correct answer from multiple choices. The numbers of correct answers are summed up; thus, the range of the diabetes knowledge score is between 0 and 11.
Time Frame: 6 month
Reporting Status: Not Posted

3. Secondary Outcome: Hypoglycaemia Awareness Score
Description: The hypoglycemia awareness questionnaire provides a score indicating the severity of hypoglycaemia unawareness. This scale ranges from 0 (maximum hypoglycaemia awareness) to 7 (minimum hypoglycaemia awareness), where a score of 4 suggests reduced hypoglycaemia awareness.
Time Frame: 6 month
Reporting Status: Not Posted

4. Secondary Outcome: Diabetes Empowerment Score (DES)
Description: Empowerment was measured by a German version of the Diabetes Empowerment Scale, a measure of diabetes-related psychosocial self-efficacy.
Time Frame: 6 month follow up
Reporting Status: Not Posted

5. Secondary Outcome: Summary of Diabetes Self-Care Activities (SDSCA)
Description: The Summary of Diabetes Self-Care Activities (SDSCA) measure is a self-report measure of diabetes self-management assessing several aspects of the diabetes regimen.
Time Frame: 6 month
Reporting Status: Not Posted

6. Secondary Outcome: Diabetes Distress Scale (DDS)
Description: Diabetes related distress was assessed by a German version of the Diabetes Distress Scale (DDS). The DDS is a 17-item self-report scale for the assessment of emotional burdens in diabetes treatment in both type 1 and type 2 diabetes.
Time Frame: 6 month follow up
Reporting Status: Not Posted

7. Secondary Outcome: CES-D Score
Description: Depressive symptoms were assessed using the German version of the Centre for Epidemiologic Studies Depression Scale (CES-D), an instrument for measuring number and severity of depressive symptoms.
Time Frame: 6 month follow up
Reporting Status: Not Posted

8. Secondary Outcome: Diabetes Self-Efficacy Scale
Description: A German version of the Diabetes Self-efficacy Scale was used to assess diabetes specific self-efficacy.
Time Frame: 6 Month Follow up
Reporting Status: Not Posted

9. Secondary Outcome: Treatment Satisfaction / Problem Areas in Dealing With Diabetes
Description: Satisfaction with current diabetes treatment was assessed by a diabetes satisfaction questionnaire developed by Kulzer et al. This questionnaire uncovers problems in dealing with diabetes, also. A high score indicates dissatisfaction with insulin therapy.
Time Frame: 6 Month Follow up
Reporting Status: Not Posted

10. Secondary Outcome: Evaluation of the Diabetes Education Course
Description: Patients satisfaction with the diabetes education programs was assessed using a self-constructed 12-item scale on specific questions regarding contents and performance of the training. Response mode was a scale ranging from 4 (apply very strong) to 0 (apply not at all). Additionally, patients were asked to give an overall grade for their course ranging from 1 (very good) to 6 (unsatisfactory).
Time Frame: 6 month Follow up
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | PRIMAS Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/79
Other Adverse Events (participants affected / at risk) | 0/81 | 0/79

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes